CLINICAL TRIAL: NCT04478825
Title: An Open Label, Proof of Mechanism Study to Explore the Efficacy and Safety of Rectally Administered BBT-401-1S in Subjects With Ulcerative Colitis
Brief Title: Efficacy and Safety of Rectally Administered BBT-401-1S in Subjects With Ulcerative Colitis
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Internal Company Decision
Sponsor: Bridge Biotherapeutics, Inc. (Industry)
Collaborators: Covance (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: BBT401-UC-004
Record Dates: First submitted 2020-07-16; First posted 2020-07-21 (Actual); Last update posted 2021-10-01 (Actual); Status verified 2021-09

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- BBT-401-1S (Experimental): BBT-401-1S, rectal administration
  Interventions: Drug: BBT-401-1S

INTERVENTIONS:
Drug: BBT-401-1S — BBT-401-1S, 8 weeks, once a day

SUMMARY:
This is an open label, single-arm, proof of mechanism study to explore the efficacy and safety of rectally administered BBT-401-1S in subjects with ulcerative colitis.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, of any race, ≥18 and ≤60 years of age on Day 1.
* Have been diagnosed with active distal UC for ≥3 months prior to Day 1, as determined by clinical and endoscopic evidence and documented in a histopathology evaluation.
* Have UC that is restricted to between the descending colon and the rectum (ie, left sided distal colitis), with demarcation of the lesion confirmed by endoscopy.
* Have a total Mayo score ≥6, an endoscopic subscore ≥2, rectal bleeding subscore ≥1, and a stool frequency subscore ≥1.

Exclusion Criteria:

* Have used any biologics or Janus kinase (JAK) inhibitors including, but not limited to, anti TNF α biologics or tofacitinib for the treatment of UC.
* Have used any purine analogues (azathioprine, mercaptopurine, or thiopurines) or immunosuppressants (methotrexate or cyclosporine) for the treatment of UC within 12 weeks or have any history of nonresponse to these medications.
* Have used any rectal therapy for the treatment of UC with exception of rectal suppository of 5-aminosalicylic acid, or any intravenous corticosteroids within 2 weeks prior to Day 1.
* Have received oral and/or rectal suppository 5-aminosalicylic acid, oral sulphasalazine, or low-dose oral corticosteroids that have been stable for <4 weeks. Doses of the drugs must remain stable until the last dose of study drug.
* Have received any other concomitant medications for UC that have been stable (ie, have not started dosing with a new drug or had a change to their dosing regimen) for <7 days or 5 half lives, whichever is longer, prior to Day 1.
* Have Crohn's disease, indeterminate colitis, ischaemic colitis, fulminant colitis, toxic megacolon, chronic pancolitis, or symptomatic intestinal stenosis.
* Have a history of extensive colonic resection (subtotal or total colectomy) or are anticipated to require surgical intervention for UC.
* Have an ileostomy or colostomy.
* Have evidence of treatment for Clostridium difficile infection or other pathogenic bowel infection within 60 days or for another intestinal pathogen within 30 days prior to Day 1.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 2 (Actual)
Dates: Start 2021-06-01 (Actual); Primary Completion 2021-08-04 (Actual); Study Completion 2021-08-24 (Actual)

PRIMARY OUTCOMES:
Endoscopic remission rate | Day 57
  measured by a Mayo endoscopic subscore of 0 or 1

SECONDARY OUTCOMES:
Endoscopic response rate | Day 57
  defined by a ≥2-point reduction from baseline in Ulcerative Colitis Endoscopic Index of Severity (UCEIS) score

OTHER OUTCOMES:
Clinical remission rate | Day 57
  measured by a total Mayo score of ≤2 points, with no individual subscore exceeding 1 point
Clinical response rate | Day 57
  measured by a reduction of ≥3 points and ≥30% improvement from baseline of total Mayo score, which includes a decrease in rectal bleeding subscore of ≥1 point or an absolute rectal bleeding subscore ≤1
Inflammatory Bowel Disease Questionnaire total score | Day 57
  measured by change from baseline. Scores for each question range between 1 and 7, reflecting poor to good health-related quality-of-life, for a range of possible total scores from 32 to 224.

CONTACTS AND LOCATIONS:
Locations (2):
- New Zealand (2):
  - P3 Research, Tauranga
  - P3 Research, Wellington